CLINICAL TRIAL: NCT04872582
Title: PD-1 Immune Checkpoint Inhibitor Combined With Bevacizumab for Patients With Metastatic Nasopharyngeal Carcinoma After Failure of Platinum-based Chemotherapy: A Single Center, Single Arm, Phase II Clinical Study.
Brief Title: Efficacy and Safety of Sintilimab Plus Bevacizumab in Metastatic Nasopharyngeal Carcinoma After Failure of Platinum-based Chemotherapy: An Open-label Phase II Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: XIANG YANQUN (Other)
Responsible Party: Sponsor-Investigator, XIANG YANQUN, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-078-01
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Nasopharyngeal Carcinoma; Chemotherapy Effect
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Bevacizumab; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 immune checkpoint inhibitor combined with bevacizumab (Experimental)
  Interventions: Drug: PD-1 Immune Checkpoint Inhibitor Combined With Bevacizumab

INTERVENTIONS:
Drug: PD-1 Immune Checkpoint Inhibitor Combined With Bevacizumab — combined
  Other Names: Sintilimab

SUMMARY:
To evaluate the efficacy and safety of PD-1 immune checkpoint inhibitor combined with bevacizumab in the treatment of metastatic nasopharyngeal carcinoma after failure of platinum-based chemotherapy.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of sintilimab combined with bevacizumab in the treatment of metastatic nasopharyngeal carcinoma (NPC) after platinum-based chemotherapy failure. The primary end point is objective response rate (ORR), the secondary end points are overall survival (OS), progression-free survival (PFS), duration of response (DOR), adverse effects and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with metastatic nasopharyngeal carcinoma are not suitable for radical local treatment.
* Previous failure of first-line platinum-containing chemotherapy (single drug or combination).
* Previously diagnosed WHO classification type II or III by histological pathology.
* At least one measurable lesion (according to RECIST1.1).
* Age between 18 and 70.
* Eastern Cooperative Oncology Group (ECOG) 0-1, and life expectation at least 3 months.
* Enough blood test.
* Participate voluntarily and sign the informed consent.

Exclusion Criteria:

* Previously diagnosed WHO classification type I by histological pathology.
* Prior exposure to anti-PD-1/PD-L1 antibodies plus anti-VEGF antibodies.
* Necrotizing lesions were found within the first 4 weeks, or the risk of massive bleeding.
* A history of interstitial pneumonia or other autoimmune diseases.
* Sever infection.
* Sever heart disease.
* HIV infection.
* Allogeneic organ transplantation
* Malignancy other than nasopharyngeal carcinoma.
* Pregnancy or breast feeding.
* Received other test drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 2 years
  The proportion of patients whose tumors shrink by a certain amount and remain in place for a certain amount of time, including complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
overall survival (OS) | 2 years
  Patients in clinical trials were randomized to the time of death from any cause
progression-free survival (PFS) | 2 years
  36/5000 The time from the commencement of a randomized clinical trial to the progression of tumorigenesis (in any respect) or death from any cause.
duration of response (DOR) | 2 years
  The time between the first assessment of a tumor as CR or PR and the first assessment of PD or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqun Xiang, Dr., Principal Investigator — Sun Yat-sen University
Locations (1):
- Yanqun Xiang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lu N, Jiang YF, Xia WX, Huang Y, Xie CM, Xu C, Ye YF, Liu GY, Bei WX, Ke LR, Li WZ, Zhang C, Wang X, Liu Q, Chen X, Chen ZX, Xie C, Liang H, Xiang YQ. Efficacy and safety of sintilimab plus bevacizumab in metastatic nasopharyngeal carcinoma after failure of platinum-based chemotherapy: an open-label phase 2 study. EClinicalMedicine. 2023 Aug 4;62:102136. doi: 10.1016/j.eclinm.2023.102136. eCollection 2023 Aug. PMID 37593221